CLINICAL TRIAL: NCT06871839
Title: The Clinical Study of Synaptic Plasticity-based Lencanumab for the Treatment of Early Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Cuibai Wei，Clinical Professor (Other)
Collaborators: Eisai (China) Pharmaceutical Co. (Unknown); Jinan Hospital, Xuanwu Hospital, Capital Medical University (Unknown); RenJi Hospital (Other); First Hospital of China Medical University (Other); Nanjing Brain Hospital (Unknown); Guangdong Provincial People's Hospital (Other); Zhejiang University (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of University of Science and Technology of China (Other); The First Hospital of Chongqing Medical University (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); West China Hospital (Other); The First Hospital of Jilin University (Other)
Responsible Party: Sponsor-Investigator, Cuibai Wei，Clinical Professor, Clinical Professor, chief physician, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: KS2024354
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer's Disease; Lecanemab; Functional Magnetic Resonance Imaging
Keywords: Alzheimer's disease; Lecanemab; functional magnetic resonance imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lecanemab treatment group: Early-stage Alzheimer's disease patients are given Lecanemab infusion treatment in conjunction with conventional anti-dementia drug therapy.
  Interventions: Drug: Lecanemab treatment group
- Conventional anti-dementia treatment: Early-stage Alzheimer's disease (AD) patients commonly take cholinesterase inhibitors such as donepezil for treatment.
  Interventions: Drug: Conventional anti-dementia treatment group

INTERVENTIONS:
Drug: Lecanemab treatment group — Lecanemab treatment group: Lecanemab Injection Concentrate Solution (active ingredient at 100 mg/mL) is provided as a sterile aqueous solution containing 100 mg/mL of Lecanemab, 50 mmol/L citric acid, 350 mmol/L arginine/arginine hydrochloride, and 0.05% (w/v) polysorbate 80, with a pH of 5.0, and each vial is capable of being drawn into a volume of 5 mL. Lecanemab is to be administered via intravenous infusion over 60 minutes in saline solution. Lecanemab must be administered using an infusion system that includes a terminal 0.22 μM inline filter. The dosage of Lecanemab is 10 mg/kg.
  All subjects in the Lecanemab treatment group receive Lecanemab infusion therapy at a frequency of once every two weeks for a continuous period of 12 months.
  Groups: Lecanemab treatment group
Drug: Conventional anti-dementia treatment group — Conventional anti-dementia treatment: Early-stage Alzheimer's disease (AD) patients routinely take cholinesterase inhibitors such as donepezil for treatment.
  Groups: Conventional anti-dementia treatment

SUMMARY:
Alzheimer's disease (AD) manifests itself in cognitive decline, impaired ability to perform daily life, and a variety of behavioral and psychiatric symptoms, seriously endangering the health of the elderly. The prevalence and disability rates of AD in China remain high, and the lack of effective treatment options has brought a heavy burden to patients and their families. Early intervention is regarded as an effective strategy to improve clinical symptoms, delay disease progression and maintain current quality of life. The humanized monoclonal antibody lencanemab (Lecanemab) was approved by the U.S. FDA in July 2023 for the treatment of mild cognitive impairment or mild dementia caused by AD, and was officially approved in January 2024 in China. Lencanemab highly targets soluble and insoluble neurotoxic β-amyloid (Aβ) proteins, reducing pathogenic Aβ plaque deposition and preventing its formation in the brains of AD patients, thus reducing neurotoxicity and improving patients' cognitive functions. In addition, lencanumab may also play a neuroprotective role by modulating synaptic plasticity and regulating neural network activity in brain neurons. However, there is a lack of clinical studies to prove this mechanism. In this study, we will enroll consecutive patients with early AD treated with lencanemab infusion as well as those receiving conventional anti-dementia therapy, and comprehensively assess the effects and intrinsic molecular mechanisms of lencanemab on synaptic function and neural networks using magnetic resonance imaging, molecular imaging positron emission tomography (PET), neuropsychological assessment, and analysis of blood cerebrospinal fluid samples.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a neurodegenerative disorder characterized by cognitive decline, impairment of daily living activities, and various behavioral and psychiatric symptoms. The most widely accepted hypothesis regarding the pathogenesis of AD is the amyloid cascade hypothesis. This hypothesis posits that the abnormal deposition of neurotoxic beta-amyloid (Aβ) is a key factor in the onset of AD. In the past two decades, anti-Aβ monoclonal antibodies aimed at reducing cerebral Aβ plaques have increasingly attracted attention in the field of AD drug development.

The humanized monoclonal antibody CAb (Lecanemab) highly targets soluble and insoluble A β[1,2] to reduce pathogenic A β plaques and prevent their formation in the brain of AD patients. Large global phase III clinical trials, including China, show that Lecanemab can slow the rate of cognitive decline in mild cognitive impairment (MCI) and mild AD within 18 months of treatment compared with placebo. However, the intrinsic mechanism by which Lecanemab delays disease progression by clearing pathogenic A β is not well understood. Previous studies have suggested that Lecanemab may have a role in improving synaptic plasticity. An animal experiment showed that the A β antibody can reverse the long-term enhanced (LTP) synaptic function defects caused by soluble A β oligomers and improve synaptic plasticity [4]. Synaptic plasticity is closely related to cognitive function. It refers to the ability to establish new connections between neurons or existing connections in the brain, which is manifested by changes in ultrastructure and functional changes of synapses, such as [5] of neurotransmitter level, neuroexcitability, electrical activity or changes in the number of postsynaptic receptors. It was shown that soluble A β oligomers are able to strongly inhibit synaptic plasticity in the normal rodent hippocampus, damage synaptic architecture, and ultimately lead to impaired cognitive [6]. Based on this, the scientific hypothesis is proposed that "Lecanemab may effectively reduce A β toxicity and protect synaptic function defects in AD brain". However, further clinical studies on the mechanism of Lecanemab on synaptic plasticity.

The purpose of this study is to prospectively evaluate the impact of continuous use of luncanemab infusion therapy on brain neural networks and synaptic plasticity in early Alzheimer's disease (AD) patients, and to explore the underlying molecular pathological mechanisms. According to the inclusion and exclusion criteria, eligible subjects are included in the screening visit period. During the screening visit, informed consent is signed, and demographic assessments are completed, along with the collection of past medical history, medication history, physical examination, and laboratory tests. Baseline neuropsychological scales, resting-state fMRI, three-dimensional structural MRI, Amyloid-PET, and blood and cerebrospinal fluid sample data are also collected. Patients are divided into a luncanemab treatment group and a conventional treatment group based on whether they receive luncanemab, and are followed up for data collection over a period of 12 months. This includes four neuropsychological assessments at 3 months, 6 months, 9 months, and 12 months of follow-up; collection of neuropsychological, resting-state fMRI, three-dimensional structural MRI, Amyloid-PET, and blood samples at baseline and at the 12-month follow-up, in accordance with patient wishes for cerebrospinal fluid sample collection; and two resting-state fMRI, three-dimensional structural MRI assessments, and blood sample collection at 6 months and 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50 and 90 years.
2. Male or female patients.
3. Patients with MCI and mild AD.
4. MMSE score ≥20, CDR overall score of 0.5 or 1.
5. Amyloid-positive confirmed by Amyloid-PET or CSF.
6. Have a reliable caregiver to accompany the patient during study visits and supervise the use of study medication during the trial.
7. Agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Patients with cognitive impairment due to reasons other than AD.
2. A history of transient ischemic attack (TIA), stroke, cerebral hemorrhage, or seizure within the 12 months prior to screening.
3. A score of >17 on the Hamilton Depression Scale at screening, or any suicidal behavior within 6 months prior to screening, at screening, or at the baseline visit, as well as any psychiatric diagnosis or symptoms that interfere with the study procedure (such as hallucinations, anxiety disorder, or paranoia).
4. Patients with a bleeding disorder or receiving anticoagulant therapy, as well as any with malignant tumors, severe gastrointestinal, kidney, liver, respiratory, immune, endocrine, and cardiovascular system diseases that affect this study.
5. A hypersensitivity reaction to ranucimab or any other ingredient in the injection solution, or to any monoclonal antibody treatment.
6. Contraindications to MRI scanning, including those with a pacemaker/defibrillator or ferromagnetic metal implants (except for skull and cardiac devices approved as safe for MRI scanning).
7. A known or suspected history of drug or alcohol abuse or dependence within the 2 years prior to screening.
8. Participation in a clinical study involving any therapeutic monoclonal antibody or novel compounds for the treatment of AD within the 6 months prior to screening, unless it can be proven that the subject was in the placebo treatment group.
9. Planning to undergo surgery requiring general anesthesia during the study period.
10. A positive pregnancy test result, lactation, or pregnancy in females at screening or baseline.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit 120 early Alzheimer's disease (AD) patients from 13 hospitals, including Xuanwu Hospital of Capital Medical University. Among them, 60 cases will be in the Lecanemab treatment group, and 60 cases in the conventional treatment group.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting-state fMRI brain network metrics (Independent Component Analysis) | 2 years
  The Lecanemab treatment group and the conventional treatment group's longitudinal changes in Independent Component Analysis (ICA) indicators after 12 months of treatment compared to baseline. ICA is a statistical technique used for extracting mutually independent signals from multivariate data, capable of measuring levels of functional connectivity within and between networks.

SECONDARY OUTCOMES:
Other resting-state fMRI brain network indicators: functional connectivity (FC) | 2 years
  Functional Connectivity (FC) is an important concept in neuroscience, primarily used to describe and analyze the interactions between different brain regions. FC is defined by measuring the similarity between brain signals from two regions.
Other resting-state fMRI brain network indicators: Granger Causality Analysis (GCA) | 2 years
  Granger Causality Analysis: Granger causality analysis is a statistical method used to analyze the causal relationships between variables.
Other resting-state fMRI brain network indicators: Spectral Dynamic Causal Model (spDCM) | 2 years
  Spectral Dynamic Causal Model (spDCM): A method for investigating the directed interactions between brain regions, also known as effective connectivity.
Rate of change in global cognition as measured by Clinical Dementia Rating (CDR) | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and conventional anti-dementia treatment using the neuropsychological scales CDR. CDR, a multidimensional scale for dementia severity, which scored 0-3, with higher scores indicating worse functioning.
Rate of change in the severity of cognitive impairment as assessed by Alzheimer's Disease Assessment Scale-Cognitive section (ADAS-cog) | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using the neuropsychological scales ADAS-cog. ADAS-cog scores range from 0-70, with higher scores indicating better global cognitive function.
Rate of change in global cognition as measured by Mini-Mental State Examination (MMSE) | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using the neuropsychological scales MMSE. MMSE scores range from 0-30, with higher scores representing better cognitive function.
Rate of change in global cognition as measured by Montreal Cognitive Assessment (MoCA) | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using the neuropsychological scales MoCA. MoCA scores range from 0-30, with higher scores representing better cognitive function.
Alzheimer's Disease Composite Score (ADCOMS) | 2 years
  ADCOMS is a weighted linear combination of selected items from three commonly used scales; it consists of 12 scoring items, with scores ranging from 0 to 1.97, where higher composite scores indicate a greater severity of the disease.
The Integrated Alzheimer's Disease Rating Scale (iADRS) | 2 years
  iADRS combines two separate scales, namely ADAS-Cog14 (scoring range from 0 to 90) and ADCS-iADL (the second part of ADCS-ADL, scoring range from 0 to 56). The total score range for iADRS is from 0 to 146, with lower scores indicating poorer performance.
Five Levels Five-Dimensional Health Scale (EQ-5D-5L) | 2 years
  The EQ-5D includes a brief descriptive system questionnaire and a visual analogue scale (EQ VAS).
  The descriptive system covers 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each of which is divided into 5 different levels to define varying degrees of difficulty: 1 = no problems; 2 = slight problems; 3 = moderate problems; 4 = severe problems; 5 = extreme problems/unable to perform. By combining the levels of each dimension, a unique health state for the subject is defined.
Alzheimer's Disease Quality of Life Scale (QOL-AD) | 2 years
  The Alzheimer's Disease Quality of Life Assessment Scale (QOL-AD), also known as the Quality of Life Assessment Scale for Senile Dementia, can evaluate multiple dimensions, including behavioral abilities, physiological functions, psychological states, interpersonal relationships, etc. The total score is the sum of the scores of 13 questions.
Rate of change in activities of daily living as assessed by Alzheimer's Disease Cooperative Study-Activity of Daily Living (ADCS-ADL) | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using the neuropsychological scales like ADCS-ADL. ADCS-ADL scores range from 0-54, with higher scores indicating better completion ability.
Rate of change in psychobehavioral symptoms as assessed by Neuropsychiatric Inventory (NPI) | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using the neuropsychological scales like NPI. Patient assessment grading scores range from 0-144 in NPI, and caregivers distress grading scores range from 0-60, with 0 representing the best.
Hamilton Anxiety Scale (HAMA) | 2 years
  Hamilton Anxiety Scale: Primarily used to assess the severity of anxiety symptoms in patients with neurosis and other disorders. The total score can be used to evaluate the severity of anxiety symptoms in patients with anxiety and depressive disorders and to assess the effects of various medications and psychological interventions. According to the data provided by the Chinese Scale Collaboration Group: a total score of ≥29 may indicate severe anxiety; ≥21 definitely indicates significant anxiety; ≥14 definitely indicates anxiety; over 7 may indicate anxiety; if less than 7, there are no anxiety symptoms.
Hamilton Depression Rating Scale (HAMD) | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using Hamilton Depression Rating Scale (HAMD):It is the most widely used scale in the clinical assessment of depressive states. The HAMD uses a 5-point rating scale for most items: (0) None, (1) Mild, (2) Moderate, (3) Severe, (4) Very Severe. A few items are rated on a 3-point scale: (0) None, (1) Mild-Moderate, (2) Severe.
  Result Analysis: <7 points are considered normal; 7-17 points are suspicious for depression; 18-24 points indicate mild or moderate depression; >24 points indicate severe depression.
Zarit Caregiver Burden Interview Scale (ZBI) | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using Zarit Caregiver Burden Interview Scale (ZBI). The score range is from 0 to 88 points, with the total score being the sum of the scores for 22 questions. The score range is from 0 to 88 points, with the total score being the sum of the scores for 22 questions.
Blood AD molecular pathology and synaptic structural protein content indicators | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using Plasma AD biomarkers (Aβ42, Aβ42/Aβ40, T-tau, P-tau181, P-tau231, P-tau217, NFL levels) and serum SV2A indicator concentration.
Cerebrospinal Fluid Synaptic Function Protein Content Assessment Indicator | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using Cerebrospinal fluid synaptic function protein content indicator (Neurotransmitter levels: Concentrations of neurotransmitters such as glutamate, acetylcholine, norepinephrine, epinephrine, dopamine, and serotonin; Neurotrophic factors: Concentration of Brain-derived Neurotrophic Factor (BDNF); Cerebrospinal fluid synaptic markers: Presynaptic Growth-associated protein 43 (GAP-43), Synaptic body-related protein 25 (SNAP25), and postsynaptic Neuronal Granulin (NRGN) markers.)
Neuroimaging biomarkers: Aβ-PET centiloid values | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using Aβ-PET centiloid values。 This is an indicator used to measure the level of amyloid deposition.

OTHER OUTCOMES:
Blood neuron-derived exosome transcriptomics-related indicators | 2 years
  Assess statistically significant difference in score between Lecanemab treatment group and Conventional anti-dementia treatment using Blood neuron-derived exosome transcriptomics-related indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Cui bai Wei, Principal Investigator — Xuan Wu Hospital of Capital Medical University
Locations (1):
- Capital Medical University Xuanwu Hospital, Beijing, China